CLINICAL TRIAL: NCT02901067
Title: STAT (STatins and Aspirin in Trauma) Trial: A Phase II, Pragmatic, Prospective, Randomized, Double-blind, Adaptive Clinical Trial Examining the Efficacy of Statins and Aspirin in the Reduction of Acute Lung Injury and Venous Thromboembolism in Patients With Fibrinolysis Shutdown
Brief Title: STAT-STatin and Aspirin in Trauma
Acronym: STAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19 pandemic and high proportion of patients meeting exclusion criteria.
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Ernest E. Moore, MD, Professor of Surgery, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COMIRB 16-0391
Record Dates: First submitted 2016-01-24; First posted 2016-09-15 (Estimated); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Wounds and Injuries; Venous Thromboembolism
Keywords: Fibrinolysis
MeSH Terms: conditions — Wounds and Injuries; Venous Thromboembolism | interventions — Aspirin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Administration of 325mg Aspirin and 20mg of Rosuvastatin mixture in a single capsule daily either orally or via a feeding tube for the duration of the patient's stay in the ICU.
  Interventions: Drug: Aspirin and Rosuvastatin
- Control (Placebo Comparator): Administration of the placebo, which is identical-looking to the Aspirin and Rosuvastatin single capsule mixture, daily either orally or via a feeding tube for the duration of the patient's stay in the ICU.
  Interventions: Drug: Placebo (for Aspirin and Rosuvastatin)

INTERVENTIONS:
Drug: Aspirin and Rosuvastatin — Patients assigned to the intervention arm will receive the standard of care anti-coagulation plus the combination experimental drugs (20mg of rosuvastatin daily and 325mg of aspirin) daily either orally or via feeding tube.
  Arms: Experimental
Drug: Placebo (for Aspirin and Rosuvastatin) — Patients assigned to the control group will receive the standard of care anti-coagulation plus identical-looking placebos either orally or via feeding tube.
  Arms: Control

SUMMARY:
This is a phase II, pragmatic, prospective, randomized, double-blind, adaptive clinical trial examining the efficacy of statins and aspirin in the reduction of acute lung injury and venous thromboembolism in patients with fibrinolysis shutdown.

DETAILED DESCRIPTION:
This protocol describes a Phase II, pragmatic, prospective, randomized, double-blind, adaptive clinical trial comparing combination rosuvastatin and aspirin therapy to placebo. Currently, there is no treatment for fibrinolysis shutdown or effective measures to prevent macro- and micro-thrombosis post-injury, thus, placebos are acceptable as the control group. Treatment for both groups would otherwise be by standard of care, which includes pharmacologic thromboembolism prophylaxis. The safety of concomitant use of VTE pharmacological prophylaxis with statins and aspirin is well documented in cardiac surgery patients.

Eligible adult patients with anticipated ICU admission will be screened for eligibility in the STAT trial (see inclusion/exclusion criteria) based on history, physical exam and clinical data obtained during their initial treatment. If deemed eligible for enrollment in the STAT trial, the patient, their legally authorized representative (LAR), or their proxy decision-maker will be contacted by our on-site professional research assistants (PRAs) for consent to enroll in the study. Only patients for whom consent is obtained within 24 hours post-injury will be eligible for randomization into the treatment phase of the study.

Upon consent, blood samples will be obtained immediately after consent at 6, 12, 24, 48, 72, 120 and 168 hours after injury. Traditional and tPA-Challenge TEG will be performed on these samples to evaluate the development of the three fibrinolysis phenotypes. Upon receiving an order for prophylactic anticoagulation, the DHMC pharmacy will randomize the patient to the control or intervention arms of the study. Randomization will occur using a computer-generated block (groups of 20 patients) random number sequence in sealed, opaque envelopes maintained at the DHMC pharmacy. Patients assigned to the intervention arm will receive the standard of care anticoagulation plus the combination experimental drugs (20mg of rosuvastatin daily and 325mg of aspirin) daily either orally or crushed via feeding tube. These doses are consistent with those currently recommended in the postoperative period following cardiac surgery. Patients assigned to the control group will receive identical-looking placebos at the same time points as the experimental group either orally or crushed via feeding tube.

Healthcare providers, PRAs and patients will be blinded to study allocation standard of care anticoagulation plus the combination placebos (produced to look and group assignment (double-blind design).

The DHMC pharmacist will be aware of the patient's treatment arm so that rapid un-blinding will be possible in the event of an adverse event possibly related to a study medication. The blood samples will be used to monitor for the type of fibrinolysis, the function of the biochemical mediators of coagulation and potential side effects of these medications, as explained in more detail below.

Study medications or placebo will be administered during ICU admission while patients are receiving the standard of care dosing of prophylactic anticoagulation (i.e. heparin or heparin-derivatives) and will be interrupted concomitantly with interruption of pharmacological VTE prophylaxis. Patients diagnosed with VTE will be withdrawn from the study drugs and will receive the appropriate VTE treatment per current ICU protocols.

The investigators will monitor function/damage of liver, renal and muscle before initiation of therapy (if the patient already has a recent test of these functions up to 12 hours prior to the initiation of therapy, the result of this test will be used to avoid unnecessary sampling), and upon the end of the therapy or as clinically necessary (i.e., any clinical indications of organ dysfunction). Stopping rules are:

1. Bleeding: Any ongoing bleeding requiring blood transfusion or operative procedure to stop bleeding. Bleeding will be monitored via monitoring of the daily measurements of hemoglobin levels, which are an integral part of the ICU protocols for trauma patients. Study medications will be unblinded and stopped if there is an unexplained drop in hemoglobin level greater than 2g/dl within 24 hours after enrollment leading to discontinuation of VTE Prophylaxis OR a drop in hemoglobin level greater than 1g/dl daily for three consecutive days leading to discontinuation of VTE Prophylaxis.
2. Liver dysfunction: Alteration in liver chemistry is a rare sequela of statin therapy. A meta-analysis of 13 placebo-controlled trials incorporating nearly 50,000 patients examined the incidence of liver toxicity (defined as elevation of hepatic transaminases greater than 3 times the upper limit of normal) in patients receiving statin therapy. 77 This study reported the incidence of elevated AST or ALT in statin-treated patients vs placebo controls as 1.14% and 1.05%, respectively (OR 1.25; 95% CI 0.99

   - 1.62). Further, the only individual drug associated with a statistically significant elevation in transaminases over a follow-up interval exceeding 3 years was fluvastatin. These and more recent data have informed expert opinion, 78 which ultimately prompted the FDA in 2012 to revoke the recommendation that liver function tests be monitored in patients taking statins. That said, given our at-risk patient population, the investigators will use the accepted definition of 3 times the baseline of the AST test as the criterion for interruption of therapy;
3. Renal dysfunction: While transient proteinuria has been observed in patients undergoing statin therapy, acute kidney injury (AKI) is a rare complication. The JUPITER randomized controlled trial incorporating approximately 17,000 patients and comparing rosuvastatin to placebo found no difference in AKI (6.0% v 5.4%; p = 0.08) between the groups. 79 In a randomized trial comparing rosuvastatin to atorvastatin, simvastatin, and pravastatin, acute renal failure was observed in 2 of 420 patients receiving high-dose rosuvastatin. 80 The AKI as serum creatinine increase greater than 2x of baseline (>Grade 1, based on AKIN criteria) as the criterion to interrupt therapy.
4. Muscle injury: Myositis and rhabdomyolysis are rare sequelae of statin therapy. A meta-analysis of 26 studies incorporating nearly 130,000 patients identified an incidence of between 1 and 4 per 10,000 patients developing rhabdomyolysis following statin therapy. 81 This meta-analysis includes a study of 12,000 patients comparing the efficacy of simvastatin 80mg with 20mg doses. In this study, the overall incidence of myolysis and rhabdomyolysis were 0.5 and 0.1 per 1000 person-years, respectively, wherein all cases of rhabdomyolysis occurred in the high dose cohort. 82 The accepted definition of myositis is muscle pain in the setting of a serum creatine kinase concentration greater than 10 times the patient's baseline.46 The investigators will use this threshold to clinically quantify myositis, preceding potential development of rhabdomyolysis, as well as the criterion to interrupt therapy.
5. If the study patient receives aspirin, as prescribed by their SICU attending, administration of the study drug will be stopped.
6. Thrombocytopenia: If the study patient's platelet count decreases below 50,000 uL requiring transfusion of platelets while receiving the study drug, administration of the study drug will be stopped. This will be monitored and recorded in our twice daily safety monitoring log.

Any of the above-mentioned stopping rules will be reported as an SAE and will trigger an immediate review by the DSMB.

ELIGIBILITY:
Inclusion Criteria: all adult trauma patients requiring admission to the surgical intensive care unit (SICU) and expected hospital stay for at least 3 days. Outside hospital transfer patients that require SICU admission less than 24 hours after their injury are also eligible for enrollment.

Exclusion criteria for prophylactic anticoagulation and for the study are:

* Known inherited bleeding disorder or coagulopathy
* Known contraindication to pharmacologic anticoagulation
* Spinal column fracture with epidural hematoma
* Head trauma/central nervous system injury

  * Severe TBI; defined as AIS Head >3
  * Intracranial hemorrhage; subdural or epidural hematoma
  * Neurosurgery service objection; neurosurgical contra-indications will be documented
* Ongoing hemorrhage requiring blood product transfusion
* Thrombocytopenia (platelet count < 50,000)
* Non-operatively managed liver or spleen injuries Grade III or above
* Known chronic kidney disease (GFR < 15ml/min)
* Rising creatinine (Cr > 1.5x baseline) at the time of enrollment
* Inclusion in any other clinical trial
* Documented previous ischemic strokes

In addition, the following exclusion criteria apply:

* Receiving statin or aspirin therapy pre-injury, as potentially being assigned for Control would increase patient's risks
* Known allergy or other contraindication to statins or aspirin
* Pregnant patients
* Prisoners, as their ability to freely consent is impaired
* Inability to obtain consent from patient or proxy prior to 48 hours post-injury
* VTE event (DVT or PE) diagnosed during current hospitalization prior to obtaining informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E Moore, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 43 patients were enrolled. Four patients withdrew after signing the consent, 2 were not randomized (1 discharged from ICU before randomization occurred, 1 received aspirin per attending prescription, making the patient ineligible for randomization).
Period: Overall Study
Arm/Group | Experimental | Control
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31.8 [23.8 to 40.6] | 39.8 [27.4 to 55] | 34.9 [26 to 45.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Mechanism of injury [Count of Participants; unit: Participants]
  Blunt | 14 | 15 | 29
  Penetrating | 5 | 3 | 8
Injury Severity Score (ISS) [Median (Inter-Quartile Range); unit: units on a scale] — The Injury Severity Score (ISS) takes values from 0 to 75, the higher the score the worse the injury. This score correlates linearly with mortality, morbidity, hospital stay and other measures of severity.
  units on a scale | 17 [14 to 26] | 22 [16 to 29] | 20 [16 to 27]
Field systolic blood pressure (SBP) [Median (Inter-Quartile Range); unit: mmHg] — Systolic blood pressure (SBP) measured in the field following the injury and before hospital arrival.
  mmHg | 101 [96 to 118] | 90 [80 to 122] | 99 [82 to 122]
Field heart rate (HR) [Median (Inter-Quartile Range); unit: beats per minute (bpm)] — Heart rate (HR) measured in the field following the injury and before hospital arrival.
  beats per minute (bpm) | 100 [87 to 116] | 98 [77 to 109] | 100 [78 to 114]
Field shock index (SI) [Median (Inter-Quartile Range); unit: units on a scale] — The shock index (SI) is an indicator of the severity of hypovolemic shock and is calculated by dividing the heart rate (HR) by systolic blood pressure (SBP). The higher the score, the worse the shock level.
  units on a scale | 1 [0.8 to 1.2] | 0.9 [0.7 to 1.1] | 1 [0.7 to 1.1]
Field Glasgow Coma Scale (GCS) [Median (Inter-Quartile Range); unit: units on a scale] — Glasgow Coma Scale (GCS) is a neurological scale which aims to give a reliable and objective way of recording the conscious state of a person for initial as well as subsequent assessment. The GCS is the summation of scores for eye, verbal, and motor responses. The minimum score is a 3 which indicates deep coma or a brain-dead state. The maximum is 15 which indicates a fully awake patient.
  units on a scale | 14 [8 to 15] | 14.5 [9 to 15] | 14 [8 to 15]
Admission lactate [Median (Inter-Quartile Range); unit: mg/dL] — Level of blood lactate measured on admission to emergency department (ED).
  mg/dL | 4.9 [3.3 to 7.9] | 5.5 [3 to 7.1] | 5 [3.3 to 7.1]
Admission pH [Median (Inter-Quartile Range); unit: units on a scale] — Level of arterial blood pH measured on admission to emergency department (ED). A normal blood pH level is 7.35 to 7.45 on a scale of 0 to 14, where 0 is the most acidic and 14 is the most basic. Trauma patients often present in acidosis.
  units on a scale | 7.3 [7.2 to 7.3] | 7.3 [7.2 to 7.3] | 7.3 [7.2 to 7.3]
Admission base excess [Median (Inter-Quartile Range); unit: mEq/L] — Level of arterial blood base excess measured on admission to emergency department (ED). Base excess refers to an excess in the amount of base present in the blood. The value is usually reported as a concentration in units of mEq/L, with positive numbers indicating an excess of base and negative a deficit. A typical reference range for base excess is -2 to +2 mEq/L.
  mEq/L | -7.2 [-12.7 to -4.3] | -8.2 [-12.8 to -3.7] | -7.8 [-12.8 to -4.3]
Admission haemoglobin [Median (Inter-Quartile Range); unit: g/dL] — First available result of haemoglobin (Hb) after admission to hospital.
  g/dL | 15 [13.1 to 15.8] | 13.1 [11.1 to 14.8] | 14.2 [12.3 to 15.3]
Admission platelet count [Median (Inter-Quartile Range); unit: 1000 cells/microL] | 266 [179 to 324] | 230.5 [169 to 305] | 239 [176 to 313]
Admission International normalized ratio (INR) [Median (Inter-Quartile Range); unit: ratio] — Defined as the first international normalized ratio (INR) obtained upon ED arrival. The international normalized ratio (INR) is an international standard for the prothrombin time (PT). This measures the time it takes for blood to clot. The normal range for a healthy person in our center is 0.83-1.19.
  ratio | 1.1 [1 to 1.3] | 1.1 [1 to 1.3] | 1.1 [1 to 1.3]
Admission partial thromboplastin time (PTT) [Median (Inter-Quartile Range); unit: seconds] | 25 [22.4 to 28.2] | 25.4 [22.7 to 27.7] | 25.3 [22.4 to 28.2]
Admission fibrinogen [Median (Inter-Quartile Range); unit: mg/dL] | 219 [218 to 236] | 179 [130 to 241] | 218 [148 to 241]
Admission D-dimer [Median (Inter-Quartile Range); unit: mcg/mL] | 5.8 [1 to 15.1] | 9 [3.9 to 20] | 9 [1.4 to 20]
Red blood cell (RBC) transfusion within first 6 hours of admission [Median (Inter-Quartile Range); unit: units] | 1 [0 to 4] | 0 [0 to 6] | 1 [0 to 4]
Fresh frozen plasma (FFP) transfusion within first 6 hours of admission [Median (Inter-Quartile Range); unit: units] | 0 [0 to 2] | 0 [0 to 5] | 0 [0 to 2]
Platelet transfusion within first 6 hours of admission [Median (Inter-Quartile Range); unit: units] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
Cryoprecipitate transfusion within first 6 hours of admission [Median (Inter-Quartile Range); unit: units] — This is the number of units of cryoprecipitate received in the first 24 hours. Most patients do not require this blood product, thus the median can be zero and the IQR can be 0 - 0 , as less than 25% of the patients required a unit of this blood product.
  units | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Massive transfusion [Count of Participants; unit: Participants] — Massive transfusion is defined as receiving 10 or more units of red blood cells (RBC) or death within 6 hours of injury and receiving 1 or more units of red blood cells.
  Participants | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence of VTE
Description: Based on screening duplex ultrasound (US) of legs and central line on day 5 or upon ICU discharge or upon symptoms of VTE (whichever comes first).
Time Frame: Day 5 or ICU discharge or upon symptoms of VTE (whichever comes first)
Measure: Number; unit: percentage of patients
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
percentage of patients | 0 | 22

2. Secondary Outcome: Fibrinolysis Phenotypes
Description: Measured by traditional and tissue plasminogen activator (tPA) - Challenge thrombelastography (TEG) lysis at 30 minutes (LY30).
Time Frame: During ICU stay at the following timepoints - 6, 12, 24, 48, 72, 120 and 168 hours
Population: We were unable to obtain samples at hour 6, as all patients were enrolled after 6 hours postinjury. The percentages below show the percentage of patients in fibrinolysis shutdown, the phenotype associated with increased risk of venous thromboembolism events.
Measure: Number; unit: percentage of patients
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
percentage of patients
  12 hours: number analyzed (Participants) | 2 | 2
  12 hours | 0 | 50
  24 hours: number analyzed (Participants) | 10 | 18
  24 hours | 43 | 57
  48 hours: number analyzed (Participants) | 16 | 16
  48 hours | 25 | 31
  72 hours: number analyzed (Participants) | 12 | 16
  72 hours | 33 | 25
  120 hours: number analyzed (Participants) | 13 | 12
  120 hours | 38 | 25
  168 hours: number analyzed (Participants) | 12 | 10
  168 hours | 33 | 20
Statistical Analysis 1: Comparison: Experimental vs Control; We hypothesized that the experimental group would present less fibrinolysis shutdown than the control group in all times measured; Test type: Superiority — This is a secondary outcome thus no power analysis was done; p > 0.05, Fisher Exact

3. Secondary Outcome: Plasminogen Activator Inhibitor (PAI) - 1 and Tissue Plasminogen Activator (tPA) Levels in Plasma
Description: To be measured in platelet poor plasma (PPP)
Time Frame: During ICU stay at the following timepoints - 6, 12, 24, 48, 72, 120 and 168 hours
Population: we were unable to measure PAI-1 and tPA in the blood samples due to lack of funding to acquire the necessary reagents and test kits. Thus, no results were produced.
Arm/Group | Experimental | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Incidence of Acute Lung Injury (ALI)
Description: Based on Berlin Criteria
Time Frame: Within two weeks post-injury
Population: Acute lung injury (ALI) was defined as by the Berlin criteria.
Measure: Number; unit: percentage of patients
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
percentage of patients | 0 | 0

5. Secondary Outcome: Ventilator Free Days
Description: As measured by ventilator-free days (VFD). VFDs are typically defined as follows (1): VFDs = 0 if subject dies within 28 days of mechanical ventilation. VFDs = 28 - x if successfully liberated from ventilation x days after initiation. VFDs = 0 if the subject is mechanically ventilated for >28 days.
Time Frame: Up to 28 days
Population: All patients had this assessment. No missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
days | 26 [23 to 28] | 26 [22 to 28]

6. Secondary Outcome: Incidence of Arterial Thrombotic Complications: Myocardial Infarction (MI) and Cerebrovascular Accident (CVA).
Description: MI and CVA were diagnosed by health care providers and documented in the EMR.
Time Frame: Up to 28 days
Population: all patients had MI and CVA work up when clinically indicated by attending in charge.
Measure: Number; unit: percentage of patients
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
percentage of patients | 0 | 0

7. Secondary Outcome: All-cause Mortality
Description: Mortality due to any cause was assessed.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p > 0.05, Fisher Exact

8. Secondary Outcome: Intensive Care Unit (ICU) Days
Description: ICU-free days will be calculated based on (28 - number of days spent in the ICU) formula
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
days | 24 [15 to 25] | 23 [15 to 26]

9. Secondary Outcome: Incidence of Multiple Organ Failure (MOF)
Description: As measured by Denver MOF score, which grades (from 0-3, with 3 indicating worst dysfunction) four organ systems (lung, kidney, liver, heart), thus varying from 0 to 12 (worst possible dysfunctions) and defines MOF as score > 3.
Time Frame: Up to 28 days
Measure: Number; unit: percentage of patients
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
percentage of patients | 0 | 0

10. Post Hoc Outcome: Pulmonary Embolism
Description: Incidence of pulmonary embolism (PE)
Time Frame: Within 30 days after injury
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
Participants | 0 | 3
Statistical Analysis 1: Comparison: Experimental vs Control; We hypothesized that the experimental group would have less pulmonary embolism events than the control group; Test type: Superiority; p = 0.10, Fisher Exact

11. Post Hoc Outcome: Incidence of Venous Thromboembolism (VTE)
Description: Includes the incidence of both deep venous thrombosis (DVT) and pulmonary embolism (PE)
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Experimental | Control
Number analyzed (Participants) | 19 | 18
percentage of patients | 0 | 22.2
Statistical Analysis 1: Comparison: Experimental vs Control; We hypothesized that the experimental group would have a lower incidence of venous thromboembolism (VTE) than the control group; Test type: Superiority; p = 0.046, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days following the injury
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 1/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/18
Other Adverse Events (participants affected / at risk) | 0/19 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=19) | Control (N=18)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastro-intestinal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=19) | Control (N=18)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — PE diagnosed 5 days after transfer out of the ICU, thus no impact on administration of study drug.
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient was diagnosed with PE on hospital day 2 and study drug discontinued per protocol.
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — PE diagnosed after transfer out of the ICU, thus no impact on administration of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02901067/Prot_SAP_001.pdf
  • Informed Consent Form (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02901067/ICF_000.pdf